CLINICAL TRIAL: NCT06471829
Title: A Phase II, Multi-site, Open-label, Dose-titration Trial to Investigate the Safety, Tolerability, Pharmacokinetics, and Efficacy of Lu AG13909 in Adults With Cushing's Disease
Brief Title: A Trial of Lu AG13909 in Adult Participants With Cushing's Disease
Acronym: BalanCeD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20433A; 2023-504733-53-00 (Other: CTIS)
Record Dates: First submitted 2024-06-18; First posted 2024-06-24 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Cushing's Disease
MeSH Terms: conditions — Pituitary ACTH Hypersecretion

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lu AG13909 (Experimental): Participants will first receive Lu AG13909 IV per predefined dosing schedule. Participants will then receive Lu AG13909 SC per predefined dosing schedule.
  Interventions: Drug: Lu AG13909

INTERVENTIONS:
Drug: Lu AG13909 — Solution for injection/infusion

SUMMARY:
This trial will evaluate the effects of Lu AG13909 in adult participants with Cushing's disease (CD). CD is a rare and serious disorder where the body makes too much of a hormone called cortisol. The main goals of this trial are to learn about

1. the effect of Lu AG13909 on cortisol levels.
2. the safety and tolerability of Lu AG13909.
3. the pharmacokinetic parameters of Lu AG13909 (how the drug is absorbed, distributed, and processed by the body).

DETAILED DESCRIPTION:
This trial is divided into 3 parts:

* Part A, consisting of 3 periods: an intravenous (IV) Titration Period, a subcutaneous (SC) Period, and a Safety Follow up Period
* Part B, consisting of 3 periods: a SC Titration Period, a Maintenance Period, and a Safety Follow-up Period
* Extension Period, consisting of a Long-Term Efficacy/Safety Period after Part B and a Safety Follow-up Period

ELIGIBILITY:
Inclusion Criteria:

* The participant is a man or woman with a confirmed diagnosis of adrenocorticotropic hormone (ACTH) driven CD of pituitary source as per current guidelines
* Morning plasma ACTH levels > lower limit of normal (LLN) and
* Evidence of a pituitary origin of the excess ACTH:

  i. Either MRI confirmation of pituitary adenoma >6 millimeters (mm), or ii. inferior petrosal sinus gradient >2, or iii. histopathology confirmation of ACTH-secreting tumour
* The participant has a 24-hour UFC >1.5 × ULN (the mean of ≥3 days of 24-hour urine collection).
* Apart from CD and associated well-controlled comorbidities (for example, diabetes mellitus and hypertension), the participant is generally healthy in the opinion of the investigator and based on medical history, physical examination, vital signs, electrocardiogram (ECG), and the results of the safety laboratory tests.
* For participants on medical treatment for hypercortisolism due to CD, pre-defined washout periods must be completed prior to the Baseline efficacy assessments.

Exclusion Criteria:

* The participant is pregnant, breastfeeding, intends to become pregnant, or is of child-bearing potential and not willing to use adequate contraceptive methods.
* The participant has a clinically significant abnormal laboratory value, ECG parameter, vital signs value, or other safety findings at the Screening Visit that indicate a potential risk to the participant's safety if enrolled, in the opinion of the investigator.
* The participant has a history of known hypersensitivity or intolerance to Lu AG13909 or its excipients.
* The participant has immediate need for pituitary surgery within 6 months from screening in the opinion of the investigator.
* The participant has severe CD per investigator judgement; among others, this could be participants with:

  i. poorly controlled hypertension ii. poorly controlled diabetes mellitus iii. severe psychiatric illness iv. compression of the optic chiasm causing any visual field defect or risk thereof v. very high risk of thromboembolic events
* The participant had pituitary surgery <3 month prior to screening.
* The participant had pituitary radiotherapy within the last 10 years.

Other protocol-defined criteria apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-06-19 (Actual); Primary Completion 2026-09-15 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Part A & Part B: Urinary Free Cortisol (UFC) Complete Response: mean UFC (mUFC) ≤ Upper Limit of Normal (ULN) at the end of the IV/SC Titration Period | Up to 490 days

SECONDARY OUTCOMES:
Number of Participants With Treatment-Emergent Adverse Events (TEAEs) | Up to 1023 days
AUC0-tau,ss: Area Under the Plasma Concentration Curve of Lu AG13909 at Steady State | Up to 1037 days
CL: Systemic Clearance of Lu AG13909 | Up to 1037 days
t½: Elimination Half-life of Lu AG13909 | Up to 1037 days
Vd: Apparent Volume of Distribution of Lu AG13909 | Up to 1037 days
SC Bioavailability (F) of Lu AG13909 | Up to 1037 days
Number of Participants With Anti-Drug Antibodies (ADAs) | Up to 1037 days
Part A Only: Cmax: Maximum Observed Plasma Concentration of Lu AG13909 | Up to 323 days
Part A Only: Tmax: Nominal Time Corresponding to the Occurrence of Cmax of Lu AG13909 | Up to 323 days
Part A & Part B: Ctrough: Minimum Observed Concentration of Lu AG13909 | Up to 659 days
Part A & Part B: Ttrough: Nominal Time Corresponding to the Occurrence of Ctrough | Up to 659 days
UFC Complete Response (mUFC ≤ ULN) or Partial Response (≥50% Reduction in UFC from Baseline and mUFC >ULN) at the End of the IV/SC Titration Period | Up to 491 days
Maintenance of UFC Complete Response (mUFC ≤ULN) at the End of the Part B Maintenance Period | Up to 337 days
Part A and Part B: Percentage Change from Baseline in mUFC at the End of the Titration Period and the Completion Visit | Baseline, up to 561 days
Part A and Part B: UFC Complete Response (mUFC ≤ ULN) or Partial Response (≥50% Reduction in UFC from Baseline and mUFC >ULN) at the Completion Visit | Up to 561 days
Part A and Part B: Late Night Salivary Cortisol (LNSC) Complete Response (Mean LNSC (mLNSC)≤ULN) or Partial Response (≥50% Reduction from Baseline in LNSC and mLNSC >ULN) at the End of the Titration Period and the Completion Visit | Up to 561 days

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — HQ_Medinfo@Lundbeck.com
Locations (23):
- France (6):
  - Centre Hospitalier Universitaire d'Angers, Angers, Cedex 09
  - Assistance Publique Hopitaux de Marseille (AP-HM) - Hopital La Conception, Marseille, Europe
  - Hopital Louis Pradel, Bron
  - APHP - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Centre Hospitalier Universitaire De Lille, Lille
  - Hopital Haut-Leveque, Pessac
- Georgia (4):
  - Ltd Tbilisi Central Hospital, Tbilisi, Europe
  - National Institute of Endocrinology, Tbilisi, Europe
  - Ltd 'Multiprofile Clinic Consilium Medulla', Tbilisi, Europe
  - Ltd Aversi Clinic, Tbilisi
- Hungary (3):
  - Semmelweis Egyetem, Belgyogyaszati es Onkologiai Klinika, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - University Hospital of Pecs, Pécs
- Italy (4):
  - Azienda Ospedale Università di Padova, Padua, Europe
  - Azienda Ospedaliero-Universitaria Pisana, Pisa, Europe
  - Azienda Ospedaliera Universitaria Sant'Andrea, Rome
  - AOU Citta della Salute e della Scienza di Torino, Torino
- Romania (3):
  - Institutul National de Endocrinologie "C.I. Parhon", Bucharest
  - Spitalul Clinic Judetean de Urgenta Cluj-Napoca, Clju-Napoca
  - Spitalul Clinic Judetean Mures, Mures
- Spain (2):
  - Hospital de la Santa Creu i de Sant Pau, Barcelona
  - Hospital Universitario Ramon y Cajal, Madrid
- University of Birmingham Institute of Metabolism and Systems Research, Birmingham, United Kingdom